CLINICAL TRIAL: NCT07093775
Title: Prognostic Implication of Tumor Grade in Patients With Node-negative Breast Cancer Aged ≤ 50 Years With 21-gene Recurrence Scores of 11-25
Brief Title: Additional Prognostic Value of Tumor Grade Beyond the 21-gene Recurrence Score
Status: Not yet recruiting | Type: Observational
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Sung Gwe Ahn, Professor, Gangnam Severance Hospital
Other Study IDs: 3-2025-0107
Record Dates: First submitted 2025-07-15; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Tumor Grade
MeSH Terms: conditions — Breast Neoplasms | interventions — vasectrin III

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tumor grade (I or II vs. III) — We compared the prognosis according to the tumor grade stratified by 21-gene recurrence score

SUMMARY:
To evaluated the prognostic significance of tumor grade in patients with node-negative, hormone receptor-positive, and human epidermal growth factor receptor 2-negative breast cancers treated according to RS-guided strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hormone receptor-positive, HER2-negative early-stage breast cancer
* Patients treated between January 2011 and December 2023
* Patients with available clinicopathologic data and 21-gene Oncotype DX assay results confirmed through electronic medical records

Exclusion Criteria:

* Patients with breast cancer under the age of 20
* Patients diagnosed with stage IV breast cancer
* Patients for whom clinicopathologic data cannot be retrieved from electronic medical records

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HR-positive, HER2-negative breast cancer who were node-negative and underwent curative surgery followed by 21-gene Oncotype DX testing
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free interval | through study completion, an average of 5 year